CLINICAL TRIAL: NCT04795154
Title: Prenatal Yoga Implementation As Complementary Therapy Of Preeclampsia Of Pregnant Woman At Puskesmas And Mandiri Practice Midwives In Palembang City
Brief Title: Prenatal Yoga as Complementary Therapy of Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. Ocktariyana, SST, M.Kes, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: OCK1982
Record Dates: First submitted 2021-01-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pre-Eclampsia
Keywords: Pre-eclampsia; Yoga; Pregnancy; exercise; complementary
MeSH Terms: conditions — Pre-Eclampsia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study was an experimental study that used pre and post-test designs in a single group. pre-group wasn't got yoga exercise, and post group was got yoga exercise was 30 minutes every 2 weeks for two months (4 times treatment). Yoga exercises technique used stretching and posture exercises (asanas) combined with deep breathing (pranayama) and meditation, to unify body, mind, and spirit (Babbar S, Parks-Savage AC, Chauhan SP, 2012). We obtained 24 samples from pregnant women> 20 weeks who had blood pressure level which was 130/80 mmHg to 140/90 mmHg got fouth times yoga exercise during pregnancy. This study was carried out in September 2020. Every each subject was measured the hypertension level by systolic and diastolic blood pressure, the protein level in urine, as well as blood platelets. The research was carried out in several public health centers where was Puskesmas Pembina and two clinics of midwives practice in Palembang city from September to November 2020.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant was pregnant women> 20 weeks who had blood pressure level which was 130/80 mmHg to 140/90 mmHg, who was approved as the subject of research and sign in the informed consent.
  The care provider was a midwife who was competent in yoga exercise, pregnancy care services, as well as competent phlebotomies.
  Investigator was the authors in this research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-test group (No Intervention): pregnant women> 20 weeks who had blood pressure level which was 130/80 mmHg to 140/90 mmHg without treatment.
- Post-test group (Experimental): pregnant women > 20 weeks who had blood pressure level which was 130/80 mmHg to 140/90 mmHg got yoga exercise, and post group was got yoga exercise was 30 minutes every 2 weeks for two months (4 times treatment). Yoga exercises technique used stretching and posture exercises (asanas) combined with deep breathing (pranayama) and meditation, to unify body, mind, and spirit (Babbar S, Parks-Savage AC, Chauhan SP, 2012).
  Interventions: Other: Yoga excercise

INTERVENTIONS:
Other: Yoga excercise — Yoga exercise in pre-eclampsia >20 weeks of pregnancy woman, treatment number was 4 times.
  Arms: Post-test group

SUMMARY:
Preeclampsia is a specific pregnancy disorder that complicates approximately 3-5% of all pregnancies. The effects on pregnant women vary from mild hypertension, severe hypertension / hypertensive crisis, eclampsia to hemolysis syndrome, elevated liver enzymes, low platelet count (HELLP), while the impact of these abnormalities on the fetus also varies from preterm birth, stunted fetal growth (CHD) to fetal death.

The initial cause of preeclampsia is still unknown, recent developments explain the molecular mechanisms behind its manifestations and especially abnormal development, placental hypoxia, endothelial dysfunction.

Prenatal yoga (yoga for pregnancy) is a modification of classical yoga which has been adapted to the physical condition of pregnant women which is done with a more gentle and slow intensity. Rakhsani A, et al., (2012) suggested that the positive effects of yoga for pregnant women are reducing occure of hypertension, preeclampsia, gestational diabetes as well as cases of intrauterine growth restriction (IUGR).

The purpose of this study was to determine the effect of prenatal yoga on reducing preeclampsia. This study was an experimental study that used pre and post-test mechanisms (paired test) with Yoga exercise treatment.

DETAILED DESCRIPTION:
Preeclampsia is a specific pregnancy disorder that complicates approximately 3-5% of all pregnancies. The effects on pregnant women vary from mild hypertension, severe hypertension / hypertensive crisis, eclampsia to hemolysis syndrome, elevated liver enzymes, low platelet count (HELLP), while the impact of these abnormalities on the fetus also varies from preterm birth, stunted fetal growth (CHD) to fetal death.

The initial cause of preeclampsia is still unknown, recent developments explain the molecular mechanisms behind its manifestations and especially abnormal development, placental hypoxia, endothelial dysfunction.

Prenatal yoga (yoga for pregnancy) is a modification of classical yoga which has been adapted to the physical condition of pregnant women which is done with a more gentle and slow intensity. Rakhsani A, et al., (2012) suggested that the positive effects of yoga for pregnant women are reducing occure of hypertension, preeclampsia, gestational diabetes as well as cases of intrauterine growth restriction (IUGR).

The purpose of this study was to determine the effect of prenatal yoga on reducing preeclampsia. This study was an experimental study that used pre and post-test mechanisms (paired test) with Yoga exercise treatment.

The number of samples wares 24 samples from pregnant women> 20 weeks who had blood pressure level which was 130/80 mmHg to 140/90 mmHg. This study was carried out in September 2020. There were three parameters to measured decreased hypertension that is blood pressure, the protein level in urine, as well as blood platelets. The research was carried out in several public health centers where was Puskesmas Pembina and two clinics of midwives practice in Palembang city from September to November 2020. Yoga exercises technique used stretching and posture exercises (asanas) combined with deep breathing (pranayama) and meditation, to unify body, mind, and spirit (Babbar S, Parks-Savage AC, Chauhan SP, 2012).

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy woman with gestational age at least 20 weeks and occurred pre-eclampsia.
* Approved as a participant with sign in an informed consent

Exclusion Criteria:

* diabetes mellitus
* kidney disorders
* heart defects
* chronic hypertension
* premature rupture of membranes
* clinical signs of infection
* Multiple pregnancies
* Death of the fetus in the womb

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Blood pressure | The blood pressure measured two times measurement that were 1 hour before yoga exercise and 1 hour after yoga exercise.
  Blood pressure is the pressure of circulating blood against the walls of blood vessels to expressed the systolic pressure (maximum pressure during on heartbeat) over diastolic pressure (minimum pressure between two heartbeats) in the cardiac cycle.
  . The blood pressure measure device used the digital sfigmomanometer.
Protein urine level | the protein urine level measured two times measurement that were 1 hour before yoga exercise and 1 hour after yoga exercise.
  The presence of proteins in urine (albumin urine) as an indication of problems in the kidneys which one is increased blood pressure. the normal value of urine albumin levels for random urine retrieval is 0-8 mg/dl. urine collected immediately after waking up which is before performing activities in the morning. about 50 ml volume of urine was measured used technique using high-performance liquid chromatography method to analysis the albumin urine.
blood platelets level | blood platelets level measured two times measurement that were 1 hour before yoga exercise and 1 hour after yoga exercise.
  Blood platelets or thrombocytes level test is count platelet level per microliter (mcL) of blood. TThe normal number of platelets in the blood is 150,000 to 400,000 platelets per microliter (mcL) or 150 to 400 × 109/L.
  the blood collected from drawing blood from a vein in the arm or hand. Obtaining a sample of blood from a vein takes a few minutes and generally causes only minimal discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Murdiningsih Murdiningsih, Principal Investigator — Politeknik Kesehatan Palembang
Locations (1):
- Poltekkes Palembang Kemenkes RI, Palembang, South of Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Babbar S, Parks-Savage AC, Chauhan SP. Yoga during pregnancy: a review. Am J Perinatol. 2012 Jun;29(6):459-64. doi: 10.1055/s-0032-1304828. Epub 2012 Mar 7. PMID 22399208
- [Result] Rakhshani A, Nagarathna R, Mhaskar R, Mhaskar A, Thomas A, Gunasheela S. The effects of yoga in prevention of pregnancy complications in high-risk pregnancies: a randomized controlled trial. Prev Med. 2012 Oct;55(4):333-340. doi: 10.1016/j.ypmed.2012.07.020. Epub 2012 Aug 2. PMID 22884667
- See also: https://pubmed.ncbi.nlm.nih.gov/22399208/ — https://pubmed.ncbi.nlm.nih.gov/22399208/